CLINICAL TRIAL: NCT04346095
Title: Comparative Analysis of Oral Sedation Versus Standard Intravenous Sedation in Vitreoretinal Surgery With Topical Anesthesia and Sub-tenon's Block
Brief Title: Oral Sedation in Vitreoretinal Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rocky Vista University, LLC (Other)
Responsible Party: Principal Investigator, Erica Podesto, OMS-II, Rocky Vista University, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0037
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Macular Holes; Intraocular Lens Opacification; Vitrectomy; Vitreous Hemorrhage; Retinal Detachment; Epiretinal Membrane; Vitreous Detachment; Intraocular Lens Dislocation
Keywords: Sedation during Vitreoretinal surgery; Oral Sedation; Anesthesia in Vitreoretinal Surgery; Oral Triazolam
MeSH Terms: conditions — Retinal Perforations; Vitreous Hemorrhage; Retinal Detachment; Epiretinal Membrane; Vitreous Detachment | interventions — Hypnotics and Sedatives; Analgesia

STUDY DESIGN:
Intervention Model Description: 1:1 randomization comparing standard procedure to experimental procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oral Sedative (Experimental): Participants will receive oral triazolam 30 minutes prior to surgery.
  Dose for BMI less than 35: 0.125 mg
  Dose for BMI greater than or equal to 35: 0.25 mg
  Followed by topical proparacaine and 6 cc sub-tenon's mixture of lidocaine and marcaine.
  Vitals will monitored by the operating room nurses.
  Interventions: Drug: Oral Sedatives with or Without Analgesia
- Intravenous Sedative (Active Comparator): This group will receive an intravenous sedative. The sedative is limited to midazolam, fentanyl, propofol.
  Follow by topical proparacaine and 6 cc sub-tenon's mixture of lidocaine and marcaine.
  IV and monitoring will be performed by anesthesiologist or CRNA.
  Interventions: Drug: Intravenous Sedatives with or Without Analgesia

INTERVENTIONS:
Drug: Oral Sedatives with or Without Analgesia — The participants will receive oral triazolam with topical proparacaine and sub-tenon's mixture of lidocaine and marcaine.
  Arms: Oral Sedative
Drug: Intravenous Sedatives with or Without Analgesia — The participants will receive intravenous midazolam, propofol or fentanyl with topical proparacaine and sub-tenon's mixture of lidocaine and marcaine.
  Arms: Intravenous Sedative

SUMMARY:
The purpose of this study is to compare the efficacy of oral sedation to intravenous sedation with anesthesiology support and monitoring.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, and providing written informed consent, a total of 40 patients will undergo vitreoretinal surgery with oral Triazolam and 40 patients will undergo vitreoretinal surgery with intravenous sedation. The IV sedative will be determined by the anesthesiologist or certified registered nurse anesthetist but limited to midazolam, propofol, and fentanyl. The study will be a prospective, cross-sectional study with a 1:1 randomized procedure and unmasked.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing vitreoretinal surgery for a variety of indications including, but not limited to, epiretinal membrane (ERM), macular hole, vitreous opacities, vitreous hemorrhage, aphakia, dislocated or displaced intraocular or crystalline lens, silicone removal, endolaser, and retinal detachment.
* American Society of Anesthesiologists rating of I-III

Exclusion Criteria:

* Undergoing vitreoretinal surgery requiring general anesthesia
* Allergy or hypersensitivity to benzodiazepines
* Pregnant or nursing females
* Previous delirium after anesthesia
* Current use of drug or alcohol on the day of surgery
* Currently on medications inhibiting cytochrome P450
* Failed anesthesia clearance
* Reported anxiety or a history of anxiolytic use
* Vitreoretinal surgery performed within the last 3 months of the current procedure
* Impaired renal or liver function

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction: scale | A patient satisfaction survey will be completed at the one-day post operative appointment.
  The patient will complete a survey at the one-day post-operative appointment. The survey consists of statements regarding the surgical procedure and experience with a scale of 1 to 6 demonstrating the patient's agreement or disagreement with the statement. Additional questions regarding the surgery and not using the 1 to 6 model will also be asked in the same survey. There will be 14 questions in the 1-6 scale portion of the survey and 4 additional questions. After all questions have been answered, the scaled questions will be analyzed for an average score out of 6 per patient. Additional questions will be analyzed by percentage of each answer. The scaled questions will be used to determine the non-inferiority of the experimental treatment. Additional questions will not be included in the non-inferiority analysis but results will be included in the study.

SECONDARY OUTCOMES:
Surgeon satisfaction: survey | The survey will be completed 10-15 minutes following the completion of the surgery.
  The surgeon will complete a survey 10-15 minutes following the completion of the surgery. The survey will include a 6 question survey with statement regarding the surgeon's experience. The surgeon will be asked to rate the statement's accuracy from a scale of 1 to 6 with 1 demonstrating strong disagreement and 6 demonstrating strong agreement. An additional yes or no question will be asked. After all questions have been answered, the scaled questions will be analyzed for an average score out of 6 per patient. Additional questions will be analyzed by percentage of each answer. The scaled questions will be used to determine the non-inferiority of the experimental treatment. Additional questions will not be included in the non-inferiority analysis but results will be included in the study.

OTHER OUTCOMES:
Anesthesiology satisfaction: survey | The survey will be completed 10-15 minutes following the completion of the surgery.
  The surgeon will complete a survey 10-15 minutes following the completion of the surgery. The survey will include a 5 question survey with statement regarding the surgeon's experience. The surgeon will be asked to rate the statement's accuracy from a scale of 1 to 6 with 1 demonstrating strong disagreement and 6 demonstrating strong agreement. An additional question will be included to the survey with a statement requiring that the participant rate the accuracy of statement with 1 representing strong agreement and 6 representing strong disagreement. After all questions have been answered, the scaled questions will be analyzed for an average score out of 6 per patient. The scaled questions will be used to determine the non-inferiority of the experimental treatment.
Registered nurse satisfaction: survey | The survey will be completed 10-15 minutes following the completion of the surgery.
  The nurse assigned to the case will complete a survey 10-15 minutes following the completion of the surgery. The survey will include a 6 question survey with a statement regarding the nurse's experience. The surgeon will be asked to rate the statement's accuracy from a scale of 1 to 6 with 1 demonstrating strong disagreement and 6 demonstrating strong agreement. An additional yes or no question will be asked. After all questions have been answered, the scaled questions will be analyzed for an average score out of 6 per patient. Additional questions will be analyzed by percentage of each answer. The scaled questions will be used to determine the non-inferiority of the experimental treatment. Additional questions will not be included in the non-inferiority analysis but results will be included in the study.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morley HR, Karagiannis A, Schultz DJ, Walker JC, Newland HS. Sedation for vitreoretinal surgery: a comparison of anaesthetist-administered midazolam and patient-controlled sedation with propofol. Anaesth Intensive Care. 2000 Feb;28(1):37-42. doi: 10.1177/0310057X0002800106. PMID 10701034
- [Background] Peeler CE, Villani CM, Fiorello MG, Lee HJ, Subramanian ML; Oral versus Intravenous Sedation Study Group. Patient Satisfaction with Oral versus Intravenous Sedation for Cataract Surgery: A Randomized Clinical Trial. Ophthalmology. 2019 Sep;126(9):1212-1218. doi: 10.1016/j.ophtha.2019.04.022. Epub 2019 Apr 16. PMID 31002834
- [Background] Rocha G, Turner C. Safety of cataract surgery under topical anesthesia with oral sedation without anesthetic monitoring. Can J Ophthalmol. 2007 Apr;42(2):288-94. PMID 17392854
- [Background] Chen M, Hill GM, Patrianakos TD, Ku ES, Chen ML. Oral diazepam versus intravenous midazolam for conscious sedation during cataract surgery performed using topical anesthesia. J Cataract Refract Surg. 2015 Feb;41(2):415-21. doi: 10.1016/j.jcrs.2014.06.027. PMID 25661136
- [Background] Donaldson M, Gizzarelli G, Chanpong B. Oral sedation: a primer on anxiolysis for the adult patient. Anesth Prog. 2007 Fall;54(3):118-28; quiz 129. doi: 10.2344/0003-3006(2007)54[118:OSAPOA]2.0.CO;2. PMID 17900211
- [Background] Dexter F, Candiotti KA. Multicenter assessment of the Iowa Satisfaction with Anesthesia Scale, an instrument that measures patient satisfaction with monitored anesthesia care. Anesth Analg. 2011 Aug;113(2):364-8. doi: 10.1213/ANE.0b013e318217f804. Epub 2011 Apr 25. PMID 21519043
- [Background] Cannon CS, Gross JG, Abramson I, Mazzei WJ, Freeman WR. Evaluation of outpatient experience with vitreoretinal surgery. Br J Ophthalmol. 1992 Feb;76(2):68-71. doi: 10.1136/bjo.76.2.68. PMID 1739718
- [Background] Carrie Chen, Daniel Luther, Thomas Acciavatti, Manju L Subramanian; Performing Ocular Procedures under Oral Sedation in Procedure Rooms: A Cost Analysis. Invest. Ophthalmol. Vis. Sci. 2019;60(9):5449. doi: https://doi.org/.